CLINICAL TRIAL: NCT04404348
Title: Cognitive Rehabilitation for Opioid Abuse-related Cognitive Impairment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted due to Covid-19 precautions
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018043
Record Dates: First submitted 2020-03-09; First posted 2020-05-27 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Three times per week for four weeks, participants will complete a computerized cognitive training session (approximately 30 minutes long).
  Interventions: Behavioral: Cognitive Training
- Control (Placebo Comparator): Three times per week for four weeks, participants will complete a computerized session (approximately 30 minutes long) that consists of inert computer games.
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Cognitive Training — Exercises used will be: Mind Bender, Divided Attention, Freeze Frame, Mixed Signals, Target Tracker, To Do List.
  Other Names: Posit Science-Brain HQ
  Arms: Intervention
Behavioral: Placebo Control — Games are drawn from the set of research control games provided by Posit Science-Brain HQ.
  Arms: Control

SUMMARY:
Research has consistently found that cognitive impairment is common in persons with a history of substance abuse. The most commonly identified impairments across all substances are in attentional and working memory functioning and executive functioning; opioid-specific research finds that memory is an additional area of common impairment. Initial research in applying cognitive rehabilitation methods to substance abuse have shown it to be helpful overall.

To develop a cognitive rehabilitation intervention that is effective for opioid abuse, this study will adapt a cognitive training program that has been shown to be effective in other patient groups. Patients in a residential opioid-abuse treatment program will undergo a cognitive evaluation and then be assigned to receive the 4-week cognitive intervention or the 4-week placebo control arm. It is expected that the intervention group will show greater gains on the cognitive post test and will have higher rated treatment adherence and opioid treatment program completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the detoxification process
* Has completed at least 8 years of formal education
* Speaks and reads English fluently
* Is beginning residential inpatient treatment for opioid abuse (note: may be receiving treatment for polysubstance abuse but opioid must be one of their regular drugs of abuse)

Exclusion Criteria:

* Unable to self-consent (has a proxy for medical decision-making, legal guardian, or been otherwise determined unable to give consent)
* Past diagnosis or suspected current diagnosis of a neurodevelopmental disorder (e.g., autism, learning disability), attention-deficit disorder, or neurocognitive disorder (e.g., dementia)
* History of major head trauma (defined as loss of consciousness for 30 minutes or longer) or brain surgery. (Note: History of concussion, including brief loss of consciousness, is okay)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mean Cognitive Change from Baseline to Endpoint | Post-intervention at week 4
  Change in overall cognitive summary score from pretest to posttest on NIH Toolbox.
Substance Abuse Program Completion Rate | Until treatment program discharge, usually 30-45 days
  Completion rate of recommended treatment program length, quantified as percentage completed

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Ford, PhD, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- 12&12, Inc, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No